CLINICAL TRIAL: NCT01857011
Title: Iron Supplementation for Acute Anemia After Postbariatric Abdominoplasty: a Randomized Controlled Trial
Brief Title: Iron Supplementation for Acute Anemia After Postbariatric Abdominoplasty
Acronym: ISAPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Juan Carlos Montano Pedroso, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISAPA UNIFESP 01
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Anemia, Iron-Deficiency; Weight Loss
Keywords: Anemia, Iron-Deficiency; bariatric surgery; abdominoplasty; surgery, plastic; iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Weight Loss | interventions — teferrol; Iron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Iron (Experimental): Intravenous Iron Sucrose 200 mg in the immediate postoperative period and first day postop.
  Interventions: Drug: Intravenous Iron sucrose
- Oral Iron (Active Comparator): Oral iron(III)-hydroxide polymaltose complex 100 mg twice daily in the fist 8 postoperative weeks.
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Intravenous Iron sucrose — Intravenous Iron Sucrose 200 mg in the immediate postoperative period and first day postop.
  Other Names: Noripurum
  Arms: IV Iron
Drug: Oral Iron — Oral iron(III)-hydroxide polymaltose complex 100 mg twice daily in the fist 8 postoperative weeks.
  Other Names: Noripurum
  Arms: Oral Iron

SUMMARY:
The purpose of this study is to determine whether intravenous or oral iron are effective in the treatment of postoperative anemia and iron deficiency in patients submitted in postbariatric abdominoplasty.

DETAILED DESCRIPTION:
Multicenter open randomized clinical trial with allocation ratio 1: 1. 56 adult patients undergoing post- bariatric abdominoplasty will be evaluated. The study group will receive 200 mg of intravenous iron in the immediate postoperative period and a second application on day 1 postoperatively. The control group will receive 100 mg of oral iron twice daily for 8 weeks. Haematological variables , iron 's profile , quality of life ( SF -36 and FACT- An) and adverse events will be assessed preoperatively and on the first , fourth and eighth weeks postoperatively .

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 a 55 years
* Prior open or laparoscopic standard limb Roux and Y gastric bypass
* BMI < 32 kg/m2
* Stability of weight loss for at least 6 months
* grade 3 abdominal deformity on the Pittsburgh scale

Exclusion Criteria:

* Illiterate
* Current smoking
* Prior IV iron use in the last 3 months
* Uncontrolled systemic diseases
* Hemoglobin < 11 g/dL
* Ferritin <11 ng/mL
* Ferritin > 100 ng/mL
* transferrin saturation <16%
* transferrin saturation> 50%
* B12 < 210 pg/mL
* Folic Acid < 3.3 ng/mL
* Albumin < 2 g/dL
* C reactive protein> 5 mg/L
* Prior Anaphylactic reaction to IV iron

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 8 postoperative weeks
  Hemoglobin level measured at 8 postoperative weeks

SECONDARY OUTCOMES:
Ferritin levels | Preoperative (one day before surgery) and 1, 4 and 8 postoperative weeks
FACIT | Preoperative (one day before surgery) and 1, 4 and 8 postoperative weeks
  The FACIT Fatigue Scale is a health related quality of life (HRQOL) questionnaire targeted to evaluate fatigue.
SF36 | Preoperative (one day before surgery) and 1, 4 and 8 postoperative weeks
  Quality of Life Questionnaire
Transferrin saturation | Preoperative (one day before surgery) and 1, 4 and 8 postoperative weeks
Hemoglobin levels | preoperative (one day before surgery) and 1, 4 postoperative weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan-Carlos Montano-Pedroso, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Montano-Pedroso JC, Bueno Garcia E, Alcantara Rodrigues de Moraes M, Francescato Veiga D, Masako Ferreira L. Intravenous iron sucrose versus oral iron administration for the postoperative treatment of post-bariatric abdominoplasty anaemia: an open-label, randomised, superiority trial in Brazil. Lancet Haematol. 2018 Jul;5(7):e310-e320. doi: 10.1016/S2352-3026(18)30071-1. PMID 29958570
- [Derived] Montano-Pedroso JC, Garcia EB, Novo NF, Veiga DF, Ferreira LM. Postoperative intravenously administered iron sucrose versus postoperative orally administered iron to treat post-bariatric abdominoplasty anaemia (ISAPA): the study protocol for a randomised controlled trial. Trials. 2016 Apr 12;17:196. doi: 10.1186/s13063-016-1300-x. PMID 27068478